CLINICAL TRIAL: NCT03178513
Title: Post-Acute Physician Home Visits: A Randomized Controlled Trial
Brief Title: Post-Acute Physician Home Visit Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jeffrey L. Schnipper, MD.,MPH., Associate Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P000719
Record Dates: First submitted 2017-06-05; First posted 2017-06-07 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: A Patient Discharged From an Acute-care Hospital Who Had an Acute Illness
MeSH Terms: interventions — House Calls

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home visit (Experimental): A participant in this arm will receive a home visit after discharge from the hospital.
  Interventions: Other: Home visit
- Usual Care (No Intervention): A participant in this arm will not receive a home visit after discharge from the hospital.

INTERVENTIONS:
Other: Home visit — The visit will be entirely patient tailored, last approximately one hour, and at a minimum will entail:
  * Medical assessment
  * Psychosocial assessment
  * Medication reconciliation
  * Follow-up of inpatient primary team's specific recommendations
  * Follow-up, as needed, with primary care team or inpatient team
  Arms: Home visit

SUMMARY:
New or worsening symptoms following discharge from the hospital likely leads to unplanned readmission. These rates are higher than desired and costly to patients, payers, and providers. Many interventions have unsuccessfully attempted to reduce readmissions, but few have provided in-home personnel to patients transitioning from acute care back to ambulatory care. Still fewer have involved a physician in the home. We therefore will test the effect of a physician home visit to a patient's home who was discharged in the last 4 days.

ELIGIBILITY:
Inclusion Criteria:

* Resides within either a 5-mile or 20-minute driving radius of Brigham and Women's Hospital (BWH) or Brigham and Women's Faulkner Hospital (BWFH) emergency room
* Has capacity to consent to study
* >=18 years old

Exclusion Criteria:

* Undomiciled
* In police custody
* Domestic violence screen positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2018-01-20 (Actual); Study Completion 2018-01-20 (Actual)

PRIMARY OUTCOMES:
New or worsening symptoms | 30 days after discharge from hospital
  "Since you got home from the hospital, have you had any symptoms at all?" If no, stop. If yes, continue.
  "I'm going to read off a list of symptoms, and I want you to tell me if that symptom is new or has gotten worse since you left the hospital. Please don't include symptoms that have stayed the same since you were in the hospital." For each affirmative, double check if the symptom is new or has gotten worse since getting out of the hospital. Only if new or worse, mark yes.

SECONDARY OUTCOMES:
Total cost, 30-days post discharge | Day of discharge to 30 days later
Total reimbursement, 30-days post discharge | Day of discharge to 30 days later
3-item Care Transition Measure, score | 30 days after discharge
Primary care provider follow-up within 14 days, y/n | Day of discharge to 14 days later
Ability to carry out the discharge plan, score | 30 days after discharge
  I would like to ask you about some more problems that you might have faced after you left the hospital one month ago. I will read some statements and ask if you agree or disagree.
Change in medication list due to home visit, y/n | Day of home visit
  Physician-initiated medication change during home visit
Receipt of prescribed medicines following discharge, y/n | 30 days after discharge
  Pharmacy confirmation
Unplanned 30-day readmission(s) after index hospitalization, y/n | 30 days after discharge
Unplanned 30-day readmission(s) after index hospitalization, # | 30 days after discharge

OTHER OUTCOMES:
Global satisfaction with care, score | 30 days after discharge
  Exploratory
Days at home since discharge, # | 30 days after discharge
  Exploratory
All-cause 30-day readmission(s) after index hospitalization, y/n | 30 days after discharge
  Exploratory
All-cause 30-day readmission(s) after index hospitalization, # | 30 days after discharge
  Exploratory
Emergency Department (ED) observation stay(s) after index hospitalization, y/n | 30 days after discharge
  Exploratory
Emergency Department (ED) observation stay(s) after index hospitalization, # | 30 days after discharge
  Exploratory
Emergency Department (ED) visit(s) after index hospitalization, # | 30 days after discharge
  Exploratory
Emergency Department (ED) visit(s) after index hospitalization, y/n | 30 days after discharge
  Exploratory
Imaging, # | 30 days after discharge
  Exploratory
Imaging, y/n | 30 days after discharge
  Exploratory
Lab orders, # | 30 days after discharge
  Exploratory
Lab orders, y/n | 30 days after discharge
  Exploratory
Physician visits, y/n | 30 days after discharge
  Exploratory
Physician visits, # | 30 days after discharge
  Exploratory
Home health utilization, days | 30 days after discharge
  Exploratory
Home health utilization, y/n | 30 days after discharge
  Exploratory
All cause 30-day mortality, y/n | 30 days after discharge
  Exploratory
Unplanned 30-day mortality, y/n | 30 days after discharge
  Exploratory
Change in medication list due to error at discharge, y/n | Visit date
  Exploratory
Pneumococcal vaccination if appropriate, y/n | 30 days after discharge
  Exploratory
Influenza vaccination if appropriate, y/n | 30 days after discharge
  Exploratory
Smoking cessation counseling if appropriate, y/n | 30 days after discharge
  Exploratory
Evaluation of ejection fraction as assessed by echocardiogram or other appropriate study, scheduled or completed, if not done within 1 year; y/n | 30 days after discharge
  Heart failure patients only; Exploratory; appropriate studies include cardiac magnetic resonance imaging, radionuclide ventriculography, single photon emission computed tomography myocardial perfusion imaging, or left ventriculography
Angiotensin converting enzyme inhibitor or angiotensin receptor blocker for heart failure with reduced ejection fraction (ejection fraction < 40%), y/n | 30 days after discharge
  Heart failure patients only; Exploratory
Beta blocker for heart failure with reduced ejection fraction (ejection fraction < 40%), y/n | 30 days after discharge
  Heart failure patients only; Exploratory
Aldosterone antagonist for heart failure with reduced ejection fraction (ejection fraction < 40%), y/n | 30 days after discharge
  Heart failure patients only; Exploratory
Lipid lowering for coronary artery disease, peripheral vascular disease, cerebrovascular accident, or diabetes, y/n | 30 days after discharge
  Heart failure patients only; Exploratory
Smoking status post-discharge | 30 days after discharge
  Heart failure patients only; Exploratory
Use of inappropriate medications in the elderly, y/n | 30 days after discharge
  Exploratory; using Screening Tool of Older Persons' potentially inappropriate Prescriptions (STOPP) and Beers criteria
Time between discharge and visit, days | Date of home visit
  Exploratory
Duration of physician visit, minutes | Date of home visit
  Exploratory

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Schnipper, MD MPH, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Brigham and Women's Faulkner Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Epstein K, Juarez E, Loya K, Gorman MJ, Singer A. Frequency of new or worsening symptoms in the posthospitalization period. J Hosp Med. 2007 Mar;2(2):58-68. doi: 10.1002/jhm.170. PMID 17431881
- [Background] Boling PA. Care transitions and home health care. Clin Geriatr Med. 2009 Feb;25(1):135-48, viii. doi: 10.1016/j.cger.2008.11.005. PMID 19217498
- [Background] Meyer GS, Gibbons RV. House calls to the elderly--a vanishing practice among physicians. N Engl J Med. 1997 Dec 18;337(25):1815-20. doi: 10.1056/NEJM199712183372507. PMID 9400040
- [Background] Wong FK, Chow SK, Chan TM, Tam SK. Comparison of effects between home visits with telephone calls and telephone calls only for transitional discharge support: a randomised controlled trial. Age Ageing. 2014 Jan;43(1):91-7. doi: 10.1093/ageing/aft123. Epub 2013 Aug 26. PMID 23978408
- [Background] Branowicki PM, Vessey JA, Graham DA, McCabe MA, Clapp AL, Blaine K, O'Neill MR, Gouthro JA, Snydeman CK, Kline NE, Chiang VW, Cannon C, Berry JG. Meta-Analysis of Clinical Trials That Evaluate the Effectiveness of Hospital-Initiated Postdischarge Interventions on Hospital Readmission. J Healthc Qual. 2017 Nov/Dec;39(6):354-366. doi: 10.1097/JHQ.0000000000000057. PMID 27631713
- [Background] Wolff JL, Meadow A, Boyd CM, Weiss CO, Leff B. Physician evaluation and management of Medicare home health patients. Med Care. 2009 Nov;47(11):1147-55. doi: 10.1097/MLR.0b013e3181b58e30. PMID 19786916